CLINICAL TRIAL: NCT02789410
Title: Intrathecal Morphine Versus Intrathecal Hydromorphone for Analgesia Following Cesarean Delivery
Brief Title: Spinal Morphine vs. Hydromorphone for Pain Control After Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Hans P. Sviggum, M.D., PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15-009421
Record Dates: First submitted 2016-05-31; First posted 2016-06-03 (Estimated); Results first posted 2019-04-25 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-03

CONDITIONS: Analgesia, Obstetrical; Obstetric Surgical Procedures
Keywords: Cesarean delivery; Analgesia; Intrathecal opioids
MeSH Terms: conditions — Agnosia | interventions — Morphine; Hydromorphone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intrathecal hydromorphone (Active Comparator): Patients will be randomized to receive a one time dose of 75 mcg intrathecal hydromorphone as part of their spinal anesthesia.
  Interventions: Drug: Hydromorphone
- Intrathecal morphine (Active Comparator): Patients will be randomized to receive a one time dose of 150 mcg intrathecal morphine as part of their spinal anesthesia.
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Morphine — Morphine is administered as part of spinal anesthesia for post-operative pain relief.
  Other Names: Duramorph
  Arms: Intrathecal morphine
Drug: Hydromorphone — Hydromorphone is administered as part of spinal anesthesia for post-operative pain relief.
  Other Names: Dilaudid
  Arms: Intrathecal hydromorphone

SUMMARY:
Intrathecal (IT) opioids are commonly administered with local anesthetic during spinal anesthesia for post-Cesarean delivery analgesia. Traditionally, IT morphine has been used but the use of IT hydromorphone is growing. A previous study has shown that the effective dose for postoperative analgesia in 90% patients (ED90) for both IT hydromorphone and IT morphine (NCT02009722). These doses were found to be 75 mcg for hydromorphone and 150 mcg for morphine. The current proposed study would compare the duration of analgesia of IT morphine vs IT hydromorphone after elective cesarean delivery. Additionally, the investigators will compare each drug with respect the incidence of nausea and pruritus.

DETAILED DESCRIPTION:
Spinal anesthesia is the most common anesthetic technique used for Cesarean delivery in the United States and across the world. Intrathecal opioids are administered with a local anesthetic during spinal anesthesia post-Cesarean delivery analgesia. The effectiveness of intrathecal morphine for post-Cesarean pain control is well established, and the use of intrathecal hydromorphone in this patient population is growing. No prospective studies have been conducted to specifically compare the efficacy of intrathecal morphine versus hydromorphone for post-Cesarean analgesia.

After intrathecal administration, opioid drug disposition depends on the lipid solubility of the individual drug. Because of its hydrophilic nature, cerebrospinal fluid (CSF) concentrations of morphine decline more slowly than similar doses of lipophilic drugs. This accounts for more rostral spread, greater dermatomal analgesia, and longer duration of action when compared to highly lipophilic opioids like fentanyl and sufentanil. When used for post-cesarean analgesia, intrathecal morphine has a duration of action between 14-36 hours with wide variation between individual patients. While hydromorphone is similar chemically to morphine, it is more lipid soluble. This decreases its spread within the intrathecal space and enhances its penetration into the dorsal horn of the spinal cord where interactions with opioid receptors occur. These differences between the two medications may influence their duration of action. Theoretically, this would reduce the duration of action of intrathecal hydromorphone when compared with intrathecal morphine. Retrospective studies have shown that the analgesic benefit for intrathecal hydromorphone appears to extend at least 12 hours after cesarean delivery and may extend up to 24 hours.

Although effective in reducing pain, intrathecal opioids are associated with side effects including pruritus, nausea, and respiratory depression. A meta-analysis reviewing twenty-eight studies which investigated intrathecal morphine versus placebo demonstrated moderate increases in the incidences of pruritus, nausea and vomiting. In fact the incidence of nausea with IT morphine has been reported to be nearly 33%. The differences in pharmacokinetics between morphine and hydromorphone may also create differences in side effect profiles. Some studies have found that hydromorphone causes less nausea and pruritus than morphine, while others have not. Although opioid-induced respiratory depression is a rare event, studies evaluating intrathecal hydromorphone for post-Cesarean delivery pain have not reported any cases of respiratory depression.

In this study, the investigators aim to compare the duration of analgesia of intrathecal morphine vs. hydromorphone for analgesia after cesarean delivery. Secondarily, the investigators will compare the side effects of each drug, including nausea and pruritus. To achieve the goals of this study, it is important to study equipotent doses of these medications. Previous work by the investigators of this study found that the effective dose for postoperative analgesia in 90% of patients (ED90) is 75 micrograms for intrathecal hydromorphone and 150 micrograms for intrathecal morphine. However, it is not known if these two equipotent medication doses provide a similar duration of analgesia.

The investigators hypothesize that 150 mcg of intrathecal morphine will result in a longer duration of analgesia when compared to 75 micrograms of intrathecal hydromorphone. Additionally, the investigators hypothesize that there will be more pruritus in the intrathecal hydromorphone group early after surgery, and no difference in side effects at 24 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status II-III women presenting for elective cesarean delivery
* Term gestation (37-42 weeks)
* Desire to have a spinal anesthesia technique for cesarean delivery

Exclusion Criteria:

* Any contraindication to the administration of a spinal technique for anesthesia
* History of intolerance or adverse reaction to opioid medications
* Chronic pain syndrome or current opioid use >30 oral morphine equivalents/day
* Allergy or intolerance to acetaminophen, ketorolac, ibuprofen, or oxycodone
* Current BMI > 50

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2016-05; Primary Completion 2017-09 (Actual); Study Completion 2018-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hans P Sviggum, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bucklin BA, Hawkins JL, Anderson JR, Ullrich FA. Obstetric anesthesia workforce survey: twenty-year update. Anesthesiology. 2005 Sep;103(3):645-53. doi: 10.1097/00000542-200509000-00030. No abstract available. PMID 16129992
- [Background] Sviggum HP, Arendt KW, Jacob AK, Niesen AD, Johnson RL, Schroeder DR, Tien M, Mantilla CB. Intrathecal Hydromorphone and Morphine for Postcesarean Delivery Analgesia: Determination of the ED90 Using a Sequential Allocation Biased-Coin Method. Anesth Analg. 2016 Sep;123(3):690-7. doi: 10.1213/ANE.0000000000001229. PMID 26974022
- [Background] Gehling M, Tryba M. Risks and side-effects of intrathecal morphine combined with spinal anaesthesia: a meta-analysis. Anaesthesia. 2009 Jun;64(6):643-51. doi: 10.1111/j.1365-2044.2008.05817.x. PMID 19462494
- [Background] Palmer CM, Emerson S, Volgoropolous D, Alves D. Dose-response relationship of intrathecal morphine for postcesarean analgesia. Anesthesiology. 1999 Feb;90(2):437-44. doi: 10.1097/00000542-199902000-00018. PMID 9952150
- [Background] Terajima K, Onodera H, Kobayashi M, Yamanaka H, Ohno T, Konuma S, Ogawa R. Efficacy of intrathecal morphine for analgesia following elective cesarean section: comparison with previous delivery. J Nippon Med Sch. 2003 Aug;70(4):327-33. doi: 10.1272/jnms.70.327. PMID 12928713
- [Background] Beatty NC, Arendt KW, Niesen AD, Wittwer ED, Jacob AK. Analgesia after Cesarean delivery: a retrospective comparison of intrathecal hydromorphone and morphine. J Clin Anesth. 2013 Aug;25(5):379-383. doi: 10.1016/j.jclinane.2013.01.014. Epub 2013 Aug 17. PMID 23965210
- [Background] Rauch E. Intrathecal hydromorphone for postoperative analgesia after cesarean delivery: a retrospective study. AANA J. 2012 Aug;80(4 Suppl):S25-32. PMID 23248827
- [Background] Rauch E. Intrathecal hydromorphone for cesarean delivery: in search of improved postoperative pain management: a case report. AANA J. 2011 Oct;79(5):427-32. PMID 23256273
- [Background] Nortcliffe SA, Shah J, Buggy DJ. Prevention of postoperative nausea and vomiting after spinal morphine for Caesarean section: comparison of cyclizine, dexamethasone and placebo. Br J Anaesth. 2003 May;90(5):665-70. doi: 10.1093/bja/aeg120. PMID 12697596
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intrathecal Hydromorphone | Intrathecal Morphine
Started | 66 | 68
Completed | 66 | 68
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intrathecal Hydromorphone | Intrathecal Morphine | Total
Number analyzed (Participants) | 66 | 68 | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.2 (4.4) | 31.9 (4.3) | 31.5 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 68 | 134
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 66 | 68 | 134

OUTCOME MEASURES:

1. Primary Outcome: NRS Score for Pain (0-10) With Movement 24 Hours After Spinal Administration
Description: Each patient will be interviewed by a member of the study team 24 hours after receiving their spinal anesthetic. Patients will be asked to rate their current level of pain on a Numeric Rating Scale (NRS) of 0 (no pain) to 10 (worst pain imaginable).
Time Frame: 24 hours after administration of spinal anesthesia
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intrathecal Hydromorphone | Intrathecal Morphine
Number analyzed (Participants) | 66 | 68
score on a scale | 4 [2.5 to 5] | 3 [2 to 4.5]
Statistical Analysis 1: Comparison: Intrathecal Hydromorphone vs Intrathecal Morphine; Test type: Superiority; p = 0.132, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Nausea
Description: The number of subjects who experienced and self-reported nausea within the first 24 hours after administration of spinal anesthesia.
Time Frame: 24 hours after administration of spinal anesthesia
Measure: Count of Participants; unit: Participants
Arm/Group | Intrathecal Hydromorphone | Intrathecal Morphine
Number analyzed (Participants) | 66 | 68
Participants | 28 | 32
Statistical Analysis 1: Comparison: Intrathecal Hydromorphone vs Intrathecal Morphine; Test type: Superiority; p = 0.590, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Pruritus
Description: The number of subjects who experienced and self-reported pruritus within the first 24 hours after administration of spinal anesthesia.
Time Frame: 24 hours after administration of spinal anesthesia
Measure: Count of Participants; unit: Participants
Arm/Group | Intrathecal Hydromorphone | Intrathecal Morphine
Number analyzed (Participants) | 66 | 68
Participants | 27 | 28
Statistical Analysis 1: Comparison: Intrathecal Hydromorphone vs Intrathecal Morphine; Test type: Superiority; p = 0.971, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Study treatment follow up was defined as 36 hours following last administration of study treatment.
Arm/Group | Intrathecal Hydromorphone | Intrathecal Morphine
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/68
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/68
Other Adverse Events (participants affected / at risk) | 0/66 | 0/68

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-21): https://cdn.clinicaltrials.gov/large-docs/10/NCT02789410/Prot_SAP_000.pdf